CLINICAL TRIAL: NCT00563004
Title: A Double-blind Placebo Controlled Study Studying the Efficacy of DBCARE in Improving Diabetes Control
Brief Title: The Effect of DBcare, a Food Supplement on Diabetes Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, pninarotman, DR, Meir Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DBcare1; DBCARE01
Record Dates: First submitted 2007-11-22; First posted 2007-11-26 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus, Non-insulin Dependant; Diabetes Mellitus Type 2; Diabetes Mellitus, on Oral Hypoglycemic Treatment; Adult Type Diabetes Mellitus
Keywords: Diabetes mellitus; Herbal treatment; Food supplement
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Patients receive the herbal medication DBCARE for 3 months
  Interventions: Dietary Supplement: DBCARE
- B (Placebo Comparator): PATIENTS RECEIVE PLACEBO PILLS
  Interventions: Dietary Supplement: DBCARE

INTERVENTIONS:
Dietary Supplement: DBCARE — Patients receive dbcare 2 tablets TID for 3 months
  Arms: A
Dietary Supplement: DBCARE — PLACEBO PILLS 2 TABLETS TID FOR 3 MONTHS
  Arms: B

SUMMARY:
DBcare is a herbal food supplement that has been used over the years in India as a "traditional"anti-diabetic formula.DBcare was not tested controlled trials in humans, yet.We intend to test the ability of DBCare to improve blood sugar level control in patients with uncontrolled diabetes.

DETAILED DESCRIPTION:
Study design: prospective, randomized, single-blind, placebo-controlled trial

Inclusion criteria:

Men and women (older than 18 years old) with type 2 diabetes and inadequate glycemic control, defined by HbA1C 8% ³ £10%.

Previous medications include any oral hypoglycemic agents, as monotherapy or in combination.

Concurrent lipid-lowering, anti-hypertensive and other medications are allowed

Exclusion criteria (before the study):

Type 1 diabetes mellitus Pregnant or lactating women Insulin treatment 3 months prior to study entry Creatinine >2 mg/dL Abnormal liver function tests GOT>X2 or GPT>X2 the upper normal limit Unstable anginal syndrome Congestive heart failure (NYHA class I-IV) Inability to follow study instructions including low compliance

Exclusion criteria (during the study):

Severe hypoglycemia (less than 50 mg%) or any hypoglycemic event requiring intravenous glucose infusion

Number of patients: 30 patients (drug) 30 patients (placebo)

Design:

Four out-patient visits, at enrollment and every month thereafter At enrollment (visit 1) physical examination will be performed and a full set of blood tests will be withdrawn At 1 week (visit 2) adjustment of hypoglycemic medications will be done and full chemistry and blood count will be taken At 6 weeks (visit 3) adjustment of hypoglycemic medications will be done and full chemistry and blood count will be taken At 12 weeks (visit 4), the end of the study, physical examination will be performed and a full set of blood tests will be withdrawn On the 2nd 3rd and 4th visits pill-count will be performed Glucose monitoring: patients will be asked to monitor fasting glucose levels at home, in the morning, on a daily basis

Drugs: identical drug containing/ placebo capsules Drugs for a month will be given in each monthly visit

Dose: 2 tablets three times daily

ELIGIBILITY:
Inclusion Criteria:

* Adults >18y
* With type 2 diabetes mellitus and inadequate glycemic control
* HBA1C >8 <10
* Previous medications include oral hypoglycemic medications,as monotherapy or in combination

Exclusion Criteria:

* Type 1 diabetes mellitus
* Pregnant or lactating women
* Insulin treatment 3 months prior to study entry
* Creatinine >2
* Abnormal liver function test GOT>2 or GPT>2 the upper limit of norm
* Unstable anginal syndrome
* Congestive heart failure NYHA 1-4
* Inability to follow study instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Reduction of more than 0.5% GBA1C in the treatment group compared to placebo | 3 months
Reduction in fasting plasma glucose of more than 20% in the treatment group compared to placebo | 3 months

SECONDARY OUTCOMES:
Reduction by half in the daily dose of oral hypoglycemic agents compared to baseline | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pnina ROTMAN-PIKELNY, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel